CLINICAL TRIAL: NCT00697047
Title: Systems of Support to Increase Colon Cancer Screening and Follow-up
Brief Title: Systems of Support (SOS) to Increase Colon Cancer Screening and Follow-up
Acronym: SOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 5R01CA121125 (NIH)
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Neoplasms; Mass Screening; Population Surveillance; Randomized controlled trial; Occult Blood; Colonoscopy; Sigmoidoscopy; Health Behavior; Colorectal Screening
MeSH Terms: conditions — Colorectal Neoplasms; Health Behavior | interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1- Usual Care (No Intervention): Usual Care (UC) includes an annual birthday letter with information on overdue screening tests including CRC screening.
- 2 - Automated Mailing (Experimental): Usual care plus automated mailing. Mailing 1 is a pamphlet about screening choices and number to call for colonoscopy. Mailing 2 is a FIT kit if not requesting colonoscopy. Mailing 3 is a Reminder letter.
  Interventions: Behavioral: Automated Mailing
- 3 - Automated Mailing Plus Assisted (Experimental): Usual care, automated mailing plus, if screening is still not completed, phone assistance by a medical assistant (MA) who asks about patients screening intent, and provides brief assistance to complete this (e.g. sends another fecal test, assists with provider order for a colonoscopy).
  Interventions: Behavioral: Automated Mailing Plus Assisted
- 4 - Auto Plus Assisted Plus Navigation (Experimental): Usual care, automated mailing, phone assistance by a medical assistant, plus navigation by a registered nurse (RN) if still not screened. Navigators are trained to use motivational interviewing techniques. They assess CRC and procedure risk, facilitate screening choice, address barriers, and provide follow-up until screening is completed.
  Interventions: Behavioral: Auto Plus Assisted Plus Navigation

INTERVENTIONS:
Behavioral: Automated Mailing — Usual Care plus Automated mailing
  Arms: 2 - Automated Mailing
Behavioral: Automated Mailing Plus Assisted — If not screened after automated mailing, MA assists with screening.
  Arms: 3 - Automated Mailing Plus Assisted
Behavioral: Auto Plus Assisted Plus Navigation — If not screened after automated mailing and assistance by MA, RN begins navigation.
  Arms: 4 - Auto Plus Assisted Plus Navigation

SUMMARY:
SOS is a four-arm randomized controlled study of ways to increase screening for colorectal cancer. About 40-50% of the people age 50 and older are not up to date on screening. This is a very important problem because screening both prevents colorectal cancer and decreases colon cancer deaths.

We are studying 3 different levels of support to help people get screened and follow-up after positive screening tests. These involve comparing to usual care stepwise increasing in intensity approaches; an automated approach of mailing information and home screening tests, this plus phone assistance by a medical assistant, both of these plus phone counseling and care management. We will also compare nurse assisted follow-up after a positive screening test compared to usual care

By doing this study we hope to increase colon cancer screening rates, and also follow-up rates for positive screening tests.

DETAILED DESCRIPTION:
Systems of Support (SOS) to Increase Colon Cancer Screening and Follow-up A. Specific Aims There is strong evidence that colorectal cancer screening (CRCS) decreases colorectal cancer (CRC) mortality and reduces colorectal cancer incidence. Despite the efficacy of screening, 40-60% of eligible adults are not screened at recommended intervals, and many have never had any type of CRCS. Screening failures occur not only from lack of screening but also from breakdowns in follow-up of positive tests, which obviates the benefits of screening. Strategies for improving the uptake of CRCS typically focus on either patients or health care providers, without describing the infrastructure changes, or systems of support (SOS), that are required to implement and sustain these changes.

We propose a two-part study using the Chronic Care Model to organize SOS. We will identify a cohort of Group Health patients aged 50 -73 years who have not had a colonoscopy (CS) in 10 years, a flexible sigmoidoscopy (FS) in 5 years, or a fecal occult blood test (FOBT) in 10 months.

Part One:

Subjects will be randomized to receive one of four interventions of stepwise increasing intensity of support.

1. Usual care (UC).
2. Automated (UC+ mailed information, access to a cancer screening hotline, mailed FOBT cards, and a reminder card).
3. Assisted (UC + automated + a medical assistant) to document screening intent and assists patients via the resources already supplied or sending requests to the patient's physician.
4. Care management (UC + automated + assisted + cancer screening nurse support) who counsels patient and assists with this screening plan (assessing procedural risk, and ordering tests).

Part Two: Patients with a positive FOBT or a positive FS (CS needed) will be randomized to one of two follow-up intervention arms: A. Usual care (which at Group Health includes a registry and physician alerts) or B. Care Management (UC + cancer screening nurse who manages care after a positive test). Our study hypotheses are that increasing levels of SOS will result in increasing CRCS rates, and care management by cancer screening nurses will increase follow-up rates after a positive test.

The primary specific aims are:

1. To compare the effectiveness of each intervention condition on increasing CRCS rates.
2. To compare the effectiveness of each intervention condition on follow-up after a positive screening test.

   The secondary aims are:
3. To assess the effects of each intervention condition on participants' cognitive, affective, and social factors related to CRCS adherence and satisfaction with medical services
4. To compare utilization, costs, and incremental cost-effectiveness of each intervention condition.

ELIGIBILITY:
Inclusion Criteria:

* Not up to date on CRCS
* Continuously enrolled in Group Health Cooperative (GHC) for 24 months
* Expected to continue to be enrolled at GHC for 24 months.

Exclusion Criteria:

* Known high risk for CRC
* History of CRC
* History of inflammatory bowel disease
* Current anticoagulation therapy
* Organ failure
* Serious illness
* Debilitating disease
* Dementia
* Nursing home resident.

Ages: 50 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4653 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Short-term adherence to CRC screening | From randomization to the end of 2 years
  To compare CRC screening adherence by randomization arm: Any screening during years 1 or 2; (b) Screening coverage during both years 1 and 2.
Long-term adherence to CRC screening | From randomization to the end of 9 years
  To compare the proportion of time participants are adherent to CRC screening long-term (initial randomization to the end of year 9).

SECONDARY OUTCOMES:
Short and long-term adherence to CRC screening for those eligible for re-randomization in year 3 | From year 3 to the end of 9 years
  To compare adherence to CRC screening, among those randomized to receive continued interventions compared to stopped interventions: a) during year 3; b) over the 7 years of follow-up from re-randomization at year 3 through the end of year 9.
Impact of SOS interventions on outcomes and CRC-related costs | From randomization to the end of 9 years
  To compare by randomization arm the impact of SOS interventions on long-term outcomes (advanced adenomas and CRC by stage), costs, and cost-effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly B Green, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data and a data dictionary without investigator support will be made available upon request to Bev.B.Green@kp.org and approval.
  The final dataset will include patient data from computerized medical records and telephone interviews with subjects. This includes demographic data (automated data and self-report), diagnoses, laboratory and procedure results and utilization data. Data will be made available as study manuscripts are published and will be de-identified prior to release for sharing.
Supporting Information: Study Protocol, ICF
Time Frame: January 1, 2021 - December 31, 2030
Access Criteria: Deidentified individual participant data and a data dictionary without investigator support will be made available upon request to Bev.B.Green@kp.org and approval.

REFERENCES:
- [Result] Meenan RT, Anderson ML, Chubak J, Vernon SW, Fuller S, Wang CY, Green BB. An economic evaluation of colorectal cancer screening in primary care practice. Am J Prev Med. 2015 Jun;48(6):714-21. doi: 10.1016/j.amepre.2014.12.016. PMID 25998922
- [Result] Green BB, Anderson ML, Wang CY, Vernon SW, Chubak J, Meenan RT, Fuller S. Results of nurse navigator follow-up after positive colorectal cancer screening test: a randomized trial. J Am Board Fam Med. 2014 Nov-Dec;27(6):789-95. doi: 10.3122/jabfm.2014.06.140125. PMID 25381076
- [Result] Green BB, Wang CY, Horner K, Catz S, Meenan RT, Vernon SW, Carrell D, Chubak J, Ko C, Laing S, Bogart A. Systems of support to increase colorectal cancer screening and follow-up rates (SOS): design, challenges, and baseline characteristics of trial participants. Contemp Clin Trials. 2010 Nov;31(6):589-603. doi: 10.1016/j.cct.2010.07.012. Epub 2010 Jul 30. PMID 20674774
- [Result] Green BB, Bogart A, Chubak J, Vernon SW, Morales LS, Meenan RT, Laing SS, Fuller S, Ko C, Wang CY. Nonparticipation in a population-based trial to increase colorectal cancer screening. Am J Prev Med. 2012 Apr;42(4):390-7. doi: 10.1016/j.amepre.2011.11.014. PMID 22424252
- [Result] Green BB, Wang CY, Anderson ML, Chubak J, Meenan RT, Vernon SW, Fuller S. An automated intervention with stepped increases in support to increase uptake of colorectal cancer screening: a randomized trial. Ann Intern Med. 2013 Mar 5;158(5 Pt 1):301-11. doi: 10.7326/0003-4819-158-5-201303050-00002. PMID 23460053
- [Result] Wang CY, de Dieu Tapsoba J, Anderson ML, Vernon SW, Chubak J, Fuller S, Green BB. Time to screening in the systems of support to increase colorectal cancer screening trial. Cancer Epidemiol Biomarkers Prev. 2014 Aug;23(8):1683-8. doi: 10.1158/1055-9965.EPI-14-0270. Epub 2014 Jun 2. PMID 24891548
- [Result] Murphy CC, Vernon SW, Haddock NM, Anderson ML, Chubak J, Green BB. Longitudinal predictors of colorectal cancer screening among participants in a randomized controlled trial. Prev Med. 2014 Sep;66:123-30. doi: 10.1016/j.ypmed.2014.06.013. Epub 2014 Jun 15. PMID 24937648
- [Result] Green BB, Anderson ML, Chubak J, Fuller S, Meenan RT, Vernon SW. Impact of continued mailed fecal tests in the patient-centered medical home: Year 3 of the Systems of Support to Increase Colon Cancer Screening and Follow-Up randomized trial. Cancer. 2016 Jan 15;122(2):312-21. doi: 10.1002/cncr.29734. Epub 2015 Oct 21. PMID 26488332
- [Result] Green BB, Anderson ML, Chubak J, Baldwin LM, Tuzzio L, Catz S, Cole A, Vernon SW. Colorectal Cancer Screening Rates Increased after Exposure to the Patient-Centered Medical Home (PCMH). J Am Board Fam Med. 2016 Mar-Apr;29(2):191-200. doi: 10.3122/jabfm.2016.02.150290. PMID 26957375
- [Derived] Green BB, Anderson ML, Cook AJ, Chubak J, Fuller S, Meenan RT, Vernon SW. A Centralized Program with Stepped Support Increases Adherence to Colorectal Cancer Screening Over 9 Years: a Randomized Trial. J Gen Intern Med. 2022 Apr;37(5):1073-1080. doi: 10.1007/s11606-021-06922-2. Epub 2021 May 28. PMID 34047921
- [Derived] Green BB, Anderson ML, Cook AJ, Chubak J, Fuller S, Kimbel KJ, Kullgren JT, Meenan RT, Vernon SW. Financial Incentives to Increase Colorectal Cancer Screening Uptake and Decrease Disparities: A Randomized Clinical Trial. JAMA Netw Open. 2019 Jul 3;2(7):e196570. doi: 10.1001/jamanetworkopen.2019.6570. PMID 31276178
- [Derived] Green BB, BlueSpruce J, Tuzzio L, Vernon SW, Aubree Shay L, Catz SL. Reasons for never and intermittent completion of colorectal cancer screening after receiving multiple rounds of mailed fecal tests. BMC Public Health. 2017 May 30;17(1):531. doi: 10.1186/s12889-017-4458-6. PMID 28558663